CLINICAL TRIAL: NCT05643300
Title: The Influence of 21st Century Skills on Clinical Decision-making in Nursing Students: a Cross-sectional Study
Brief Title: 21st Century Skills of Nursing Students
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Seyma Demir, Research Assistant Doctor (PhD), Abant Izzet Baysal University
Other Study IDs: AIBU-HSF-SDEMIR-03
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Students; Nurse's Role
Keywords: Students, Nursing; Clinical Decision-Making; 21st-century skills
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Data collection from participants via questionnaire

SUMMARY:
It was aimed to investigate the effect of Twenty first century (21st) century skills on the clinical decision making of nursing students. Within the scope of the cross sectional study, answers to the following research questions will be sought:

* What are the 21st century skill levels of nursing students?
* Are nursing students' 21st century skills affected by their sociodemographic characteristics?
* What are the clinical decision-making levels of nursing students?
* Are the clinical decision-making levels of nursing students affected by their sociodemographic characteristics?
* Do nursing students' 21st century skills affect their decision-making levels?

DETAILED DESCRIPTION:
In this cross-sectional study, it is planned to investigate the effects of 21st century skills on clinical decision making of nursing students. Junior and senior students of a nursing undergraduate program in Turkey will be recruited. The universe of the research consists of junior (167 people) and senior (210 people) nursing students of a nursing undergraduate program in a university in Turkey in the 2022-2023 academic year. Sample selection will not be made and those who volunteer to participate will be included. According to the university's nursing program curriculum, first and second year students were excluded from the study because they did not have clinical practice experience. Data will be collected using an Information Form containing sociodemographic data, Multidimensional 21st Century Skills Scale and Nursing Decision Making Instrument. Data collection forms will be collected on the online platform in line with the link created through Google forms. The link address will be shared via students' smartphones. After explaining to the students that the purpose of the study before the application, the participation is on a voluntary basis and the confidentiality of the information obtained will be ensured, they will be asked to fill in the online questionnaire by entering the address in the link. Data collection time is planned to take approximately 10-15 minutes. The dependent variable of the study was clinical decision making; independent variables are 21st century skills and sociodemographic characteristics. In this direction, data analysis will be based on the comparison of dependent and independent variables. If the data is continuous, it will be displayed as percentile, mean, standard deviation; comparison will be made by correlation analysis. Discrete data will be compared with dependent variable according to data level by t test or analysis of variance. The effect of 21st century skills and sociodemographic characteristics of nursing students on clinical decision making will be tested with multivariate regression analysis enter method. For categorical variables, a dummy model will be created and converted into continuous data. Statistical significance value will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Nursing undergraduate program junior and senior students
* Volunteering to participate

Exclusion Criteria:

* Nursing undergraduate program 1st and 2nd year students

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of junior and senior of the undergraduate nursing program. Students in lower grades do not have any clinical experience due to the curriculum of the program. Therefore, clinical decision-making is best measured by recruiting junior and senior students.
Sampling Method: Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
21st century skills (questionnaire) | Baseline
  It will be measured by the Multidimensional 21st Century Skills Scale. It is a 5-point Likert-type scale (ranging from 1-Strongly Disagree to 5-Strongly Agree) consisting of 41 items and five sub-dimensions: Knowledge and technology literacy skills, critical thinking and problem solving skills, entrepreneurship and innovation skills, social responsibility and leadership skills, career consciousness. Scores range from 41 to 205, and the higher the scores, the higher the 21st century skill levels.The Cronbach's Alpha coefficient of the Turkish scale is 0.86 and the coefficient of each sub-dimension is over 0.70.
Clinical decision making (questionnaire) | Baseline
  It will be measured by the Nursing Decision Making Instrument. The Turkish scale has 24 items and one dimension. Five-point Likert type is evaluated as "never or almost never-1 to almost always-5". Even numbered items reflect intuitive decision making, odd numbered items reflect analytical decision making.The scores that can be obtained from the scale vary between 24-120. A score over 67 is considered analytical, a score between 68-78 is considered semi-rational, and a score over 78 is considered intuitive decision making. As the scores obtained from the scale decrease, it is concluded that the participants make more analytical decisions, and as the scores increase, they make more intuitive decisions. The Cronbach's Alpha coefficient of the Turkish scale is 0.97.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyma Demir Erbaş, PhD, Principal Investigator — Bolu Abant Izzet Baysal University, Faculty of Health Sciences
Locations (1):
- Bolu Abant Izzet Baysal University Faculty of Health Sciences, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No